CLINICAL TRIAL: NCT02588209
Title: Cognitive Screening and Cognitive Training in Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGK11-52
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMART Training (Experimental): This group will receive the Strategic Memory Advanced Reasoning Training (SMART) program, twice a week for four weeks.
  Interventions: Behavioral: Strategic Memory Advanced Reasoning Training
- Health (Active Comparator): This group will receive the Brain Health Workshop educational program, twice a week for four weeks.
  Interventions: Behavioral: Brain Health Workshop

INTERVENTIONS:
Behavioral: Strategic Memory Advanced Reasoning Training — SMART teaches strategies to improve the ability to process information.
  Other Names: SMART
  Arms: SMART Training
Behavioral: Brain Health Workshop — Brain Health Workshop provides information about brain health in a seminar format. Topics include: sleep, nutrition, and exercise.
  Arms: Health

SUMMARY:
This study will provide cognitive screenings for seniors age 50 and older. It will also investigate the benefits of two different cognitive training programs for seniors who have lower baseline performance on memory and/or gist reasoning tests.

DETAILED DESCRIPTION:
This study consists of two parts which includes cognitive screening and cognitive training. Participants will initially participate in the cognitive screening portion of the study. If qualified, participants will participate in the cognitive training portion of this study which includes additional cognitive communication, neuropsychological testing, and EEG.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive complaints in the absence of dementia
* Participate in tasks involving motor abilities such as use of at least one arm and hand
* Read, speak, and comprehend English
* At least 50 years of age
* Comprehend simple instructions, perform tasks, and take part in intervention

Exclusion Criteria:

* Not proficient in reading,comprehending, and speaking English
* History of learning disability, stroke, cognitive impairment, major psychiatric illness, alcoholism, or substance abuse

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Improvement in memory or thinking after brain training | beginning (0 weeks) to end (4 weeks)
  To examine short-term effects of treatment on cognition using neuropsychological measures

SECONDARY OUTCOMES:
Measures changes in brain wave activity | beginning (0 weeks) and end (4 weeks)
  Electrophysiological responses will be recorded using event related potential to monitor responses to yes/no stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Chapman, PhD, Principal Investigator — Center for Brain Health, University of Texas at Dallas
Locations (1):
- UTD Center for BrainHealth, Dallas, Texas, United States

REFERENCES:
- [Derived] Mudar RA, Nguyen LT, Eroh J, Chiang HS, Rackley A, Chapman SB. Event-related neural oscillation changes following reasoning training in individuals with Mild Cognitive Impairment. Brain Res. 2019 Feb 1;1704:229-240. doi: 10.1016/j.brainres.2018.10.017. Epub 2018 Oct 17. PMID 30342001